CLINICAL TRIAL: NCT01954433
Title: Costs and Consequences of Three Common Orthopedic Procedures on the Upper Extremity - Health Economic Investigation (Cost-effectiveness and Cost-utility Analyses) With Before and After Surgery Comparison
Brief Title: Costs and Consequences of Three Common Orthopedic Procedures on the Upper Extremity
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Collaborators: Winterthur Institute of Health Economics (WIG), Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: CUA-OrthopaedicsOE-CIP-v2.0
Record Dates: First submitted 2013-09-17; First posted 2013-10-01 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Degenerative Arthritis of Left Glenohumeral Joint; Degenerative Arthritis of Right Glenohumeral Joint; Rotator Cuff Tear Arthropathy; Rotator Cuff Tear; Trapeziometacarpal Osteoarthritis
Keywords: Cost-effectiveness analyses; Cost-utility analyses; Upper extremity; Orthopedic; Shoulder arthroplasty; Rotator cuff tear repair; Resection interposition suspension arthroplasty
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Operated TSA Patients: Patients with glenohumeral arthritis and/or rotator cuff tear arthropathy who were operated and received a total shoulder prosthesis
  Interventions: Procedure: Operated TSA Patients
- Non-operated TSA Patients: TSA-patients, indicated for treatment with a total shoulder prosthesis, who decided not to operate
- Operated RCR Patients: Patients with rotator cuff tear who were operated and received a rotator cuff reconstruction by arthroscopy
  Interventions: Procedure: Operated RCR Patients
- Non-operated RCR Patients: RCR-patients, indicated for rotator cuff reconstruction by arthroscopy, who decided not to operate
- Operated TMC OA Patients: Patients with trapeziometacarpal (TMC) osteoarthritis who were operated and received a resection interposition suspension arthroplasty of the TMC joint
  Interventions: Procedure: Resection interposition suspension arthroplasty (RISA)
- Non-operated TMC OA Patients: TMC OA-patients, indicated for surgical treatment (resection interposition suspension arthroplasty), who decided not to operate

INTERVENTIONS:
Procedure: Operated TSA Patients — Total shoulder prosthesis: Anatomic or reverse total shoulder replacement is a well-standardized procedure usually performed under general anesthesia with the patient in a beach-chair position
  Groups: Operated TSA Patients
Procedure: Operated RCR Patients — Arthroscopic rotator cuff tear reconstruction. The shoulder arthroscopy is performed according to internal and international standard procedure with patients positioned in beach-chair position under general anesthesia.
  Groups: Operated RCR Patients
Procedure: Resection interposition suspension arthroplasty (RISA) — One of five surgical techniques can be used in this study, as routinely performed by each surgeon:
  1. RISA with FCR-Ligament (flexor carpi radialis ligament) modified according to Epping
  2. RISA with FCR-Ligament modified according to Weilby
  3. RISA with APL-Ligament (abductor pollicis longus ligament)
  4. RISA with Graftjacket modified according to Weilby
  5. Resection arthroplasty
  Groups: Operated TMC OA Patients

SUMMARY:
This study compares costs and effectiveness / utility of three common orthopedic surgeries in shoulder and hand from the perspective of the Swiss health system and the clinic.

The cost of health care is continuously rising, making economic considerations part of the decision process, in particular for the allocation of available resources. However, cost-effectiveness and cost-utility studies of interventions in the upper extremities are rare. The purpose of this study is to gain more information and to provide a basis for the decision process.

DETAILED DESCRIPTION:
Among various recognized methods used to assess the benefits and value of medical services, cost-effectiveness analysis (CEA) and cost-utility analysis (CUA) are taking an increasingly important role. Over recent years, economic evaluations gained interest in orthopedics, suggesting the inclusion of economic factors in addition to traditional outcome measures in the evaluation of surgical interventions.

This is a prospective mono-center observational study involving three independent patient groups (Total shoulder prosthesis for arthritis (TSA), Arthroscopic repair of rotator cuff tears (RCR), Trapeziectomy for Trapeziometacarpal Osteoarthritis (TMC OA)) of 150 patients each. Before-and-after comparisons will be made: Cost-effectiveness and cost-utility data collected post-operatively up to one (TMC OA) and two years (TSA and RCR) will be compared with those collected up to one year pre-operatively. Eligible patients unwilling to receive surgery will be followed-up for one and two years, respectively, to allow for a parallel comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient aged 18 years and over
* Patient willing and able to give written informed consent to participate in the study including all pre-surgical and post-surgical follow-up examinations
* Patient authorizing that their health insurance be contacted to provide health-related costs for the purpose of this study

Specific inclusion Criteria:

TSA:

* patients diagnosed with primary or secondary glenohumeral arthritis and/or rotator cuff tear arthropathy
* indicated for treatment with a total anatomic or reverse shoulder prosthesis or

RCR:

* patients diagnosed with partial or complete rotator cuff tear
* indicated for rotator cuff reconstruction by arthroscopy

or

TMC OA:

* patients diagnosed with TMC OA
* indicated for surgical treatment by resection interposition suspension arthroplasty of the TMC joint

Exclusion Criteria:

* General medical contraindication to surgery
* Revision operations
* Known hypersensitivity to the materials used
* Tumour / malignoma
* Addiction or other disorders (e.g. neuromuscular, psychiatric or metabolic disorder) that would preclude accurate evaluation
* Recent history of substance abuse
* Legal incompetence
* Pregnant women
* Participation in any other medical device or medicinal product study within the previous months that could influence the results of the present study

Specific exclusion Criteria:

* Other joints operated in the same session, except arthrodesis of the metacarpophalangeal (MCP) I joint
* Patients with rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with shoulder arthritis and/or rotator cuff tear arthropathy indicated for total shoulder prosthesis (TSA)
  * Patients with rotator cuff tear indicated for arthroscopic rotator cuff reconstruction (RCR)
  * Trapeziometacarpal osteoarthritis (TMC OA) patients indicated for resection interposition suspension arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness and cost-utility of the targeted interventions | Change from 1 year before OP at 1 (TMC OA) or 2 (RCR, TSA) years post OP (/ after enrollment for non-operated patients)
  To calculate the cost-effectiveness and cost-utility of the targeted interventions we will assess the following parameters before and after surgery:
  * Health-related costs which include all direct and indirect costs before and after surgery (productivity via work status/salary and Work Productivity and Activity Impairment Questionnaire WPAI)
  * Quality-Adjusted Life years (QALYs)
  * Incremental Cost Effectiveness Ratio (ICER)
Change in quality of life | preOP, immediately preOP, 2 weeks, 3, 6, 12 months postOP respectively 6 and 12 months after enrollment for non-operated patients
  Quality of life (utilities) derived using EuroQoL EQ-5D-5L. The primary analysis will investigate the change between immediately before and one year after surgery.

SECONDARY OUTCOMES:
Change in quality of life in TSA- and RCR-Patients after 2 years | 2 years postOP (/ after enrollment for non-operated patients)
  Quality of life (utilities) derived using EQ-5D-5L
Complications | From enrollment up to 1 or 2 years after surgery
  Patient-level risk of intervention-related complications (during non-operative management, intra-operative, post-operative including events leading to revision surgeries).
Local imaging Parameters (assessed from MRT, ultrasound, radiographs) | TSA: preOP, 6 months, 1 and 2 years postOP, RCR: preOP, 6 months postOP, TMC OA: preOP
  TSA preOP:
  * Status of the rotator cuff (intact / partial rupture)
  * Supraspinatus muscle atrophy
  * Amount of fatty infiltration in the rotator cuff muscles
  * Acromiohumeral distance
  * Severity of arthrosis
  TSA postOP:
  * Head position with respect to glenoid
  * Occurrence of osteolysis and migration
  * Cortical bone resorption (when a shaft is implanted)
  * Status of the Tuberculum Majus
  RCR preOP:
  * Location and extent of the injury of the rotator cuff (partial / complete rupture)
  * Amount of fatty infiltration in the rotator cuff muscles
  * Extend of tendon retraction
  * Signs of tendon degeneration
  RCR postOP:
  * Position of the anchors
  * Postoperative tissue growth
  TMC OA preOP:
  * Stage of Osteoarthritis
  * Occurrence of articular chondrocalcinosis
  * Involvement of the scapho-trapezio-trapezoidal (STT) joint
  * Distance between the scaphoid and the metacarpal
Change of Constant (Murley) score (CS) due to surgery in TSA- and RCR-patients | preOP, immediately preOP, 3, 6 months postOP. TSA additionally: 12, 24 months postOP
  The Constant (Murley) score is possibly the most commonly used tool for assessment of shoulder function. The physician asks and documents answers to Quality of life questions (pain and activity of daily living, ability to work, sleep, sports and leisure) and certain clinical parameters (active range of motion, abduction strength). The different scales will be summed and normalized to 0 = worst to 100 = best. A German version is available for clinical use.
  With the CS we can assess the change and gain in functional shoulder outcome.
Change of range of motion due to surgery in TSA- and RCR-patients | preOP, immediately preOP, 3, 6 months postOP. TSA additionally: 12, 24 months postOP
  Additional to th Constant score we assess the
  * passive abduction
  * passive elevation
  * active and passive external rotation by 0°
  * active and passive external-internal rotation by 90°
Change of Kapandji index and grip + key pinch strength due to surgery in TMC OA-patients | preOP, immediately preOP, 3, 6, 12 months postOP
  The ability to oppose the thumb of both hands will be quantified using the Kapandji index. The flexion/extension of the metacarpo-phalangeal (MCP) and inter-phalangeal (IP) joint of the affected and contralateral thumb will be measured with an electrical Goniometer (ELINK, Biometrics Ltd., Gwent, UK).
  Grip strength as well as key pinch strength of both hands will be measured with the help of an electrical dynamometer and pinch gauge (ELINK, Biometrics Ltd., Gwent, UK). Three records will be taken and the mean value will be taken for analyses. The standardized testing position as recommended by the American Society of Hand Therapists will be used.
Change of Shoulder Pain and Disability Index (SPADI) during study participation in TSA-patients | preOP, immediately preOP, 3, 6, 12, 24 months postOP; respectively 6, 12 and 24 months after enrollment for non-operated patients
  The Shoulder Pain and Disability Index (SPADI) is a short, self-administered questionnaire that provides an item scoring by a visual analogue scale (VAS) from 0 (no pain/no difficulty, i.e. best) to 11 (worst pain imaginable/so difficult required help, i.e. worst). Five items assess pain and 8 items disability of the arm (function). The unweighted means of the 5 pain and the 8 function items will be transformed into the scale from 0 (=worst) to 100 (=best) for both scales and are used to determine pain and function scores. The average of these two scores then gives the total SPADI score. A validated German version is available.
Change in Oxford Shoulder Score (OSS) during study participation in RCR-patients | preOP, immediately preOP, 3, 6, 12 and 24 months postOP; respectively 6, 12 and 24 months after enrollment for non-operated patients
  The OSS is a condition-specific questionnaire developed for patients with a degenerative or inflammatory state of the shoulder. It contains 12 items to be answered by the patient independently, which deal with pain (degree, time point) and possible handicaps in private and professional life. There are five categories of response for every question, corresponding to a score ranging from 0 to 4. Scores are combined to give a single score, with a range from 0 (worst outcome) to 48 (best outcome). The score can also be standardized from 0 to 100 (best) for comparison with other outcome instruments. A German version of this questionnaire is available and it is suitable for patient-based outcome after rotator cuff repair.
Change in Michigan Hand Outcomes Questionnaire (brief MHQ) during study participation in TMC OA-patients | preOP, immediately preOP, 3, 6, 12 months postOP; respectively 6 and 12 months after enrollment for non-operated patients
  The Michigan Hand Outcomes Questionnaire MHQ was specifically designed to measure health state domains important to patients with hand disorders. In contrast to the widely applied DASH, the MHQ seems to be more sensitive to functional changes in hand patients. Compared to the DASH and Patient Evaluation Measure, the MHQ shows the highest correlation in finger patients with grip strength and range of motion.
  In this study we will use a short version of the MHQ that includes only 12 questions for patients with acute or chronic disorders of the hand. The answers are rated on a 5-point Likert scale and scores are normalized on a scale of 0 to 100. The brief MHQ demonstrated an excellent test-retest reliability.
Change in Disability of the Arm, Shoulder and Hand questionnaire (QuickDASH) during study participation in TSA- and TMC OA-patients | TMC OA + TSA: preOP, immediately preOP, 3, 6, 12 months postOP. TSA additionally: 24 months. 6, 12 and 24 months after enrollment for non-operated patients.
  The Disability of the Arm, Shoulder and Hand questionnaire (DASH) is a comprehensive self-administered questionnaire about symptoms and functioning of the entire upper extremity. The DASH enquires about the ability to perform simple and complex activities of daily living (ADL) that are commonly performed with either one or both arms. The total score is derived from the unweighted mean of 30 items, of which at least 27 have to be answered. The QuickDASH is a more efficient version of the DASH outcome measure that appears to retain its measurement properties. It contains eleven items and is similar with regard to scores and properties to the full DASH. A validated full-length German version is available that can be used in the shortened version.
Change in Subjective shoulder value (SVV) during study participation in TSA- and RCR-patients | RCR + TSA: preOP, immediately preOP, 3, 6, 12, 24 months postOP; respectively 6, 12 and 24 months after enrollment for non-operated patients
  The Subjective Shoulder Value (SSV) is based on a single question that is answered subjectively by the patients. The formulation of this question is: "What is the overall percent value of your shoulder if a completely normal shoulder represents 100%?" It is an easily administered measure of shoulder function.
Change in general health during study participation | preOP, immediately preOP, 3, 6, 12 months postOP. TSA + RCR additionally: 24 months postOP; ; respectively 6, 12 and 24 months after enrollment for non-operated patients
  The outcome measure "general health" is a composite of these three questions:
  * patients will be asked to report their general health status on a visual analog scale from 0 (worst possible health) to 100 (best possible health) using the EQ-5D-5L instrument.
  * In addition, patients will be asked to assess their current state of health related to the operated shoulder or hand at follow-up compared to the state before surgery. This so-called 'transition' question has the possible answers 'much worse', 'slightly worse', 'equal', 'slightly better', and 'much better'.
  * A similar question will be asked regarding their perceived change in quality of life at follow-up compared to the state before surgery.
Change in level of satisfaction during study participation | preOP, immediately preOP, 3, 6, 12 months postOP. TSA + RCR additionally: 24 months postOP. ; 6, 12 and 24 months after enrollment for non-operated patients
  The outcome measure "level of satisfaction" is a composite of these two questions:
  * Patients are asked to rate their level of satisfaction, with the help of a numeric rating scale (NRS: 0-10), in terms of how the outcome met up to their preoperative expectations.
  * Finally, they will be asked whether - with their current knowledge of the outcome - they would again choose the operation if they found themselves in similar circumstances to those which prevailed preoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias P Flury, Dr. med., Principal Investigator — Schulthess Klinik; Laurent Audigé, DVM PhD, Study Director — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

REFERENCES:
- [Derived] Marks M, Grobet C, Audige L. Validity, responsiveness and minimal important change of the EQ-5D-5L in patients after rotator cuff repair, shoulder arthroplasty or thumb carpometacarpal arthroplasty. Qual Life Res. 2021 Oct;30(10):2973-2982. doi: 10.1007/s11136-021-02849-7. Epub 2021 May 10. PMID 33973108
- See also: Schulthess Klinik — http://www.schulthessklinik.ch